CLINICAL TRIAL: NCT01204905
Title: Raltegravir and Maraviroc in Combination for the Treatment of Antiretroviral Naïve HIV-1 Infected Patients
Brief Title: R5 Integrase Study in HIV-1 Naive Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HP-00045769
Record Dates: First submitted 2010-09-16; First posted 2010-09-17 (Estimated); Results first posted 2018-10-18 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: HIV Infections
Keywords: HIV-1; CD4; Viral Load; Human Immunodeficiency Virus (HIV)
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Raltegravir Potassium; Maraviroc

STUDY DESIGN:
Intervention Model Description: Single arm treatment study
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Open Label ART (Experimental): Patients received raltegravir 400 mg PO BID and maraviroc 300 mg PO BID in combination for 48 weeks.
  Interventions: Drug: Raltegravir and Maraviroc in combination

INTERVENTIONS:
Drug: Raltegravir and Maraviroc in combination — Raltegravir 400 mg tablet twice a day, ~12 hours (10 to 14 hours) apart
  Maraviroc 300 mg tablet twice a day, ~12 hours (10 to 14 hours) apart
  Other Names: Raltegravir (Isentress); Maraviroc(Selzentry)

SUMMARY:
This is a pilot, open-label study of raltegravir and maraviroc in combination for the treatment of antiretroviral naïve patients. The study will enroll 7 antiretroviral naïve patients with CD4 counts ≥ 350 and viral loads > 5,000. The subjects will be followed for 48 weeks. The combination of these two agents has the potential to be a potent regimen with minimal metabolic complications. However, they have not been studied in combination previously.

This pilot study proposes to evaluate this combination in antiretroviral naïve patients to document the safety and efficacy of this combination in order to provide clinicians with a treatment regimen that minimizes the risk of metabolic complications.

DETAILED DESCRIPTION:
Seven antiretroviral naïve HIV infected participants will be treated with a combination of raltegravir and maraviroc and followed for 48 weeks to determine the time to virologic suppression of (HIV-1 viral load < 50 copies/ml).

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection
* CD4 count ≥ 350
* RNA > 5,000
* CCR5 tropic virus
* Baseline genotype without significant mutations known to confer antiretroviral drug resistance to currently licensed antiretroviral agents
* Antiretroviral naïve (< 7 days of experience)
* 18-75 years of age
* Subject able to provide informed consent for the study
* Women of child-bearing age agree to remain abstinent or use (or have their partner use) an acceptable method of birth control throughout the study. Acceptable method of birth control is defined as intrauterine device (IUD), diaphragm with spermicide, contraceptive sponge, condom, vasectomy.

Exclusion Criteria:

* Dual/mixed tropic virus,
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >2.5 times the upper limits of normal;
* Total bilirubin >1.5 mg/dL,
* Women pregnant or breastfeeding,
* History of malignancy
* Enrollment in an experimental protocol with concomitant use of drugs known to impact or be impacted in terms of pk or drug-drug interactions with either raltegravir or maraviroc. This includes inducers of UGT1A1 ( such as rifampin, phenytoin, Phenobarbital rifabutin, St. John's wart) as well as CYP3A inhibitors (such as ketoconazole, itraconazole, clarithromycin , nefazodone and telithromycin) and CYP3A inducers (such as rifampin, carbamazepine, Phenobarbital and phenytoin)
* Enrollment in an experimental protocol having received investigational agents(antiretroviral or non-antiretroviral) within 30 days of study enrollment
* Chronic active hepatitis B infection
* Subject has a history or current evidence of any condition, therapy, laboratory abnormality or other circumstance that might confound the results of the study, or interfere with the patient's participation for the full duration of the study, such that it is not in the best interest of the patient to participate.
* Subject is unlikely to adhere to the study procedures, keep appointments, or is planning to relocate during the study.
* Subject requires or is anticipated to require any of the prohibited medications noted in the protocol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2010-09; Primary Completion 2014-05-16 (Actual); Study Completion 2014-05-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert R. Redfield, MD, Principal Investigator — University of Maryland, Institute of Human Virology
Locations (1):
- University of Maryland, Institute of Human Virology, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Open Label ART: Patients received raltegravir 400 mg PO BID and maraviroc 300 mg PO BID in combination for 48 weeks.
  Raltegravir and Maraviroc in combination: Raltegravir 400 mg tablet twice a day, ~12 hours (10 to 14 hours) apart
  Maraviroc 300 mg tablet twice a day, ~12 hours (10 to 14 hours) apart
Period: Overall Study
Arm/Group | Open Label ART
Started | 7
Completed | 5
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Open Label ART
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 40 [26 to 61]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Viral Load
Description: Percentage of subjects with HIV-1 viral load < 50 copies/ml
Time Frame: 48 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label ART
Number analyzed (Participants) | 7
Participants | 4
Statistical Analysis 1: Comparison: Open Label ART; Test type: Other — This was a pilot study with a small sample population. There were no power calculations performed; The percentage of patients with HIV-1 viral loads less than 50 c/ml at 48 weeks

2. Secondary Outcome: Viral Suppression
Description: Time to attainment of virologic suppression
Time Frame: 48 weeks
Measure: Number; unit: weeks
Arm/Group | Open Label ART
Number analyzed (Participants) | 7
weeks | 6
Statistical Analysis 1: Comparison: Open Label ART; Test type: Other — There were no power calculations performed due to the size of the pilot study; Number of weeks to virologic suppression

ADVERSE EVENTS:
Time Frame: 48 weeks
Arm/Group | Open Label ART
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 2/7
Other Adverse Events (participants affected / at risk) | 6/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label ART (N=7)
Thrombocytopenia (Cardiac disorders) | 1 (1) — Not study related, Adverse Event occurred before study drug started.
Gunshot Wound (Gastrointestinal disorders) | 1 (1) — Not study related
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label ART (N=7)
Fatigue (General disorders) | 1 (1) — Fatigue resolved
Light headedness (General disorders) | 1 (1) — Resolved
Mouth ulcers (General disorders) | 1 (1) — Resolved
Dental Infection (Infections and infestations) | 1 (1) — Treatment Resolved
Syncopal Episode (General disorders) | 1 (1) — Dehydration, resolved
Kidney Stones (Renal and urinary disorders) | 1 (1) — Treatment resolved

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes